CLINICAL TRIAL: NCT03746223
Title: Combined Intravitreal Methotrexate and R2 Regimen Followed by Lenalidomide Maintenance in Newly-diagnosed Primary Vitreoretinal Lymphoma
Brief Title: Intravitreal Methotrexate and R2(Rituximab & Lenalidomide) Regimen in Newly-diagnosed Primary Vitreoretinal Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-003
Record Dates: First submitted 2018-11-06; First posted 2018-11-19 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2018-11

CONDITIONS: Primary Intraocular Lymphoma
Keywords: intravitreal methotrexate injection; rituximab; lenalidomide; Primary vitreoretinal lymphoma
MeSH Terms: conditions — Intraocular Lymphoma | interventions — Methotrexate; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R2-R/IV-MTX（methotrexate） (Experimental): experimental arm will be treated rituximab plus lenalidomide (R2) regimen for 6 cycles and followed by lenalidomide maintenance for 2 years, meanwhile intravitreal methotrexate will be given as protocol
  Interventions: Drug: Methotrexate; Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Methotrexate — 400ug intravitreal injection every week for 4 doses in the induction phase, every 2 weeks for 2 doses as consolidation, then every month for 10 doses as maintenance
Drug: Rituximab — Rituximab：375mg/m2 intravenous infusion d1, every 28 days for 1 cycle. 6 cycles will be prescribed as protocol
Drug: Lenalidomide — 25mg Qd, oral , d1-21 in 28-day cycle in the induction phase and maintenance phase.

SUMMARY:
This is a prospective single arm phase II study, and the purpose of this study is to evaluate the efficiency of R2 regimen (rituximab & lenalidomide) combined with intravitreal methotrexate and followed by lenalidomide maintenance in newly-diagnosed primary intraocular lymphoma. Progression free survival (PFS) of the cohort is the primary endpoint.

DETAILED DESCRIPTION:
All the patients will be treated with R2 regimen （Rituximab 375mg/m2 IV d1, lenalidomide 25mg d1-21, 28 days per cycle) as induction regimen, meanwhile intravitreal methotrexate was given at a dose of 400ug for 16 doses.

The response will be evaluated every 3 cycles. After 3 Cycles, patients who achieved complete remission (CR) or partial remission (PR) will receive 3 more cycles of R2 regimen. The patients with stable disease (SD) or progressed disease (PD) will withdraw from the trial and receive salvage regimens. After total 6 induction cycles, the investigators evaluate the efficiency again, the patients with CR or PR will go to lenalidomide maintenance for 2 years or until progression of the disease (PD), unacceptable toxicity, or patient/investigator discretion. And the patients with SD or PD will receive salvage regimen.

During following-up, surveillance ophthalmologic examination and brain magnetic resonance imaging (MRI) scans can be performed every 3 months up to the first 2 years, followed by doctor visit every 6 months up to 5 years or the disease relapses.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed primary vitreoretinal lymphoma
* ECOG≤2
* creatinine clearance rate (CCR) ≥ 60ml/h, according to Cockcroft-Gault
* Total bilirubin < 2 upper limits of normal, alanine aminotransferase（ALT） < 3 upper limits of normal
* Sign the Informed consent
* Women of childbearing potential must understand that the study medication could have a potential teratogenic risk. They should undergo complete contraception during the study period.
* Male subjects must agree to use condoms throughout study drug therapy.

Exclusion Criteria:

* primary central nervous system lymphoma involved eyes and brain
* systemic B cell lymphoma involved eyes
* Pre-existing uncontrolled active infection
* Clinical evidence of grade 3 or 4 heart failure as defined by the New York Heart Association criteria
* Pregnancy or active lactation
* Co-existing tumors
* HIV（human immunodeficiency virus） or HBV（hepatitis B virus） or HCV（hepatitis C virus） infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
2 years progression-free survival | from the date of treatment to the subject finished his 2 years follow-up phase or the disease relapsed or the death due to lymphoma
  2 years progression-free survival was calculated from the date of therapy until death from lymphoma or 2-year follow-up without relapsing

SECONDARY OUTCOMES:
overall response rate(ORR) | 4 weeks after the end of 6 cycles of induction (each cycle is 28 days).
  ORR was calculated by the proportion of patients who achieved complete remission and partial remission.

CONTACTS AND LOCATIONS:
Overall Officials: Daobin Zhou, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Zhang X, Zou D, Yin J, Zhang L, Wang X, Jia C, Wang W, Zhao D, Zhou D, Zhang W, Zhang M. Lenalidomide and Rituximab Regimen Combined With Intravitreal Methotrexate Followed by Lenalidomide Maintenance for Primary Vitreoretinal Lymphoma: A Prospective Phase II Study. Front Oncol. 2021 Jun 24;11:701507. doi: 10.3389/fonc.2021.701507. eCollection 2021. PMID 34249763